CLINICAL TRIAL: NCT07116278
Title: Deriving Candidate Diagnostic and Prognostic Network Biomarkers for Chronic Pain Using the QuantalX DELPHI TMS-EEG System
Brief Title: TMS-EEG Biomarkers for Chronic Pain
Acronym: DELPHI TMS-EEG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-40427
Record Dates: First submitted 2025-07-10; First posted 2025-08-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: pain; chronic pain; fibromyalgia
MeSH Terms: conditions — Chronic Pain; Pain; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Longitudinal TMS-EEG (Other): Each visit will involve completion of the TMS-EEG intervention.
  Interventions: Device: QuantalX DELPHI-MD (TMS-EEG)

INTERVENTIONS:
Device: QuantalX DELPHI-MD (TMS-EEG) — Direct Electro-Physiological Imaging medical device (DELPHI-MD), developed by QuantalX Neuroscience, is a neurophysiological assessment system which utilizes a specific TMS-EEG protocol that automatically analyzes specific features of this brain response to reproduce numerical output measures. DELPHI-MD has previously shown to differentiate different healthy age groups, mild dementia and Parkinson's Disease (PD) from age matched healthy control. In addition, DELPHI-MD measures are correlated to white matter microstructural differences in post stroke and TBI patients. This multimodal approach allows for the evaluation of several neurophysiological mechanisms such as cortical reactivity, excitation and inhibition in local and distal regions, effective connectivity, and neural plasticity, characterized as modifications that outlast the stimulation period. The investigators predict that Delphi-MD has the potential to identify features of brain function altered in pain syndromes.

SUMMARY:
In this study the investigators aim to assess the correlates of neurophysiological measures (measurement of brain magnetically evoked response) using DELPHI system. The DELPHI system device is a computerized, electromechanical medical device that produces and delivers non-invasive Transcranial Magnetic Stimulation (TMS) fields to induce electrical currents directed at regions of the cerebral cortex and records the resultant Electroencephalogram (EEG) brain electrophysiological response. DELPHI analyzes the TMS Evoked Potential (TEP) and produces quantitative output measures.

Objectives include:

* To use TMS-evoked EEG measures of brain function in patients with chronic pain using the QuantalX DELPHI system to predict patient specific pain diagnoses using machine learning classification methods.
* To evaluate longitudinal associations between TMS-evoked EEG measures and ratings of chronic pain.
* To monitor associations between TMS-evoked EEG biomarkers and therapy success for three different classes of medications.

DETAILED DESCRIPTION:
Chronic pain is the leading cause of disability worldwide. Patients with chronic pain have highly variable responses to available treatments, leading to trial-and-error based interventions that delay relief, prolong suffering, and increase reliance on potentially addictive opioid analgesics. This hallmark variability between individual patients is a key barrier to the development of reliable biomarkers for diagnosis and treatment selection. Chronic pain is associated with maladaptive reorganization of brain circuits involved in sensory, emotional, and cognitive aspects of pain. However, specific abnormalities and their relationships to personalized outcomes are unknown. Here, the investigators propose to collect measures of brain network connectivity, excitability, and plasticity using the QuantalX DELPHI-MD (TMS-EEG) system to identify mechanistic biomarkers for patient diagnosis and treatment prognosis. This is a prospective, pilot cohort study. Relationships uncovered during analysis of pilot data will be used to support future experimental research and better characterize specific measures that may be useful to collect in ongoing patient outcome research at UCSF.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18-80 with a diagnosis of chronic pain agreeing to participate in all study procedures. To maximize accrual and phenotypic variability in the sample for planned analyses, we include patients meeting ICD-11 criteria for chronic pain, a duration-based parent code for several common, clinically relevant pain conditions. Patients must have pain lasting more than 6 months.

Exclusion Criteria:

* Neurologic disorders: Dementia, Severe neurocognitive disorder (MoCA < 22), Severe aphasia, Seizure disorder, certain structural brain lesions (e.g., intracranial mass lesions, neoplasms, hydrocephalus, sequelae of meningitis, MS plaques), cerebral palsy, or complete paralysis
* Major psychiatric disorders (e.g., Bipolar Disorder, Schizophrenia), suicidal thoughts
* Subjects with any metallic brain implant or fragments (such as shunt, pacemaker, clips, coils, bullet fragments, cochlear implants).
* Subjects with any implanted devices activated or controlled by physiological signals and/or ferromagnetic or other magnetic sensitive metals implanted in the head or anywhere within 12 inches/30 cm from the stimulation coil.
* Subjects using medications that may alter electroencephalography (EEG) waveforms, including ketamine and benzodiazepines, are eligible to participate, but will be asked to hold these medications 4-8 hours prior to the study visits, as appropriate.
* Pregnant or breastfeeding woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
TMS-Evoked Potential Amplitude | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  The QuantalX DELPHI (TMS-EEG) system will be used to generate N45 potential amplitudes from the primary motor cortex. The DELPHI System is used for acquisition of physiological signals of Electroencephalography (EEG) from the scalp in response to magnetic stimulation. It consists of a DELPHI amplifier, a computer (workstation), a patient EEG cap, a transcranial magnetic stimulation (TMS) device and "Figure 8" stimulation coil. To limit the effect of medications on EEG results, participants will be asked to hold medications known to significantly alter EEG waveforms (including ketamine and benzodiazepines) 4-8 hours prior to the study visits, as appropriate. The device can also generate a range of regional and global metrics of brain excitability (e.g., N100 potential amplitudes), plasticity (e.g., change in N45 amplitude after conditioning pulses), and connectivity (e.g., between region coherence) at each scheduled clinic visit.
Visual analog scores (VAS) | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  Real time pain intensity and unpleasantness ratings from 0 to 100.

SECONDARY OUTCOMES:
Numerical Rating Scales (NRS) | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  Real time pain intensity and unpleasantness ratings from 1 to 10.
Pain Body Maps | Visit 1(Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  A validated visual representation of the human body allowing patients to record the location and severity of pain.
NIH PROMIS questionnaires | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  The NIH PROMIS toolbox contains a host of survey questions tailored to measurement of specific disease states such as pain, global health and function. We will specifically use the Global Health, nociceptive and neuropathic pain (short forms), pain interference (short form), and Patient global impression of change.
McGill Pain Questionnaire (MPQ) | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  The McGill Pain Questionnaire is a validated measure of multiple domains of pain processing, including sensory and affective pain processing as well as nociceptive and neuropathic pain. Scores range from 0-45 with higher scores indicating more pain.
Pain Catastrophizing Scale (PCS) | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  Validated scale measuring emotional responses to pain to track pain-related symptoms. Scores range from 0-52 with higher scores indicating higher pain catastrophizing.
Beck Depression Inventory-II (BDI-II) | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  Validated measure of clinical depression symptoms to quantify and track mood over time. Scores range from 0-63 with higher scores indicating more depression.
World Health Organization Disability Assessment Schedule (WHODAS) | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  Assessment of functional disability from the WHO to track level of function over time. Scores range from 0-100 with higher scores indicating more disability.
Pittsburgh Sleep Quality Index (PSQI) | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  Validated scale that measures sleep and insomnia symptoms. Scores range from 0-21 with higher scores indicating worse sleep quality.

OTHER OUTCOMES:
Thermal Pain Detection Threshold | Visit 1 (Baseline), Visit 2 (1-3 months after the first visit), Visit 3 (3-6 months), Visit 4 (6-9 months), Visit 5 (9-12 months)
  Cold pain and heat pain (°C) thresholds are assessed using Quantitative Sensory Testing (QST) .

CONTACTS AND LOCATIONS:
Overall Officials: Julian Motzkin, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified TMS-EEG data with our industry collaborators. We will share de-identified TMS-EEG, QST, and self-reported pain data via open science repositories.
Supporting Information: Study Protocol, Analytic Code
Time Frame: All data will be deposited to OpenNeuro and OSF within 6 months of the final publication resulting from these data.
Access Criteria: To request access of the data, researchers will use the standard processes at OSF, which involve contacting the study author for use permission. Data can be accessed freely on UCSF MyResearch.

REFERENCES:
- [Background] Zifman N, Levy-Lamdan O, Suzin G, Efrati S, Tanne D, Fogel H, Dolev I. Introducing a Novel Approach for Evaluation and Monitoring of Brain Health Across Life Span Using Direct Non-invasive Brain Network Electrophysiology. Front Aging Neurosci. 2019 Sep 9;11:248. doi: 10.3389/fnagi.2019.00248. eCollection 2019. PMID 31551761
- [Background] Maidan I, Zifman N, Hausdorff JM, Giladi N, Levy-Lamdan O, Mirelman A. A multimodal approach using TMS and EEG reveals neurophysiological changes in Parkinson's disease. Parkinsonism Relat Disord. 2021 Aug;89:28-33. doi: 10.1016/j.parkreldis.2021.06.018. Epub 2021 Jun 29. PMID 34216938
- [Background] Levy-Lamdan O, Zifman N, Sasson E, Efrati S, Hack DC, Tanne D, Dolev I, Fogel H. Evaluation of White Matter Integrity Utilizing the DELPHI (TMS-EEG) System. Front Neurosci. 2020 Dec 21;14:589107. doi: 10.3389/fnins.2020.589107. eCollection 2020. PMID 33408607
- [Background] Fogel H, Levy-Lamdan O, Zifman N, Hiller T, Efrati S, Suzin G, Hack DC, Dolev I, Tanne D. Brain Network Integrity Changes in Subjective Cognitive Decline: A Possible Physiological Biomarker of Dementia. Front Neurol. 2021 Aug 30;12:699014. doi: 10.3389/fneur.2021.699014. eCollection 2021. PMID 34526957